CLINICAL TRIAL: NCT04604145
Title: Evaluation of Self-Collected Saliva Samples Without Viral Transport Media for SARS-CoV-2 Testing Via RT-PCR
Brief Title: Self-Collected Saliva Samples Without Viral Transport Media for COVID-19 Testing Via RT-PCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nolan Hudson, Research Associate/Medical Technologist, Principal Investigator, David Grant U.S. Air Force Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FWH20200198H
Record Dates: First submitted 2020-10-23; First posted 2020-10-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV Infection; Polymerase Chain Reaction; Laboratory Testing
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive NP results (Other): SARS-CoV-2 testing on self-collected saliva specimens, associated with a positive NP result, using the Eppendorf Thermal Cycler Polymerase chain reaction (PCR) system
  Interventions: Diagnostic Test: SARS-CoV-2 testing on the Eppendorf Thermal Cycler PCR system using self-collected saliva as the specimen
- Negative NP results (Other): SARS-CoV-2 testing on self-collected saliva specimens, associated with a negative NP result, using the Eppendorf Thermal Cycler Polymerase chain reaction (PCR) system
  Interventions: Diagnostic Test: SARS-CoV-2 testing on the Eppendorf Thermal Cycler PCR system using self-collected saliva as the specimen

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 testing on the Eppendorf Thermal Cycler PCR system using self-collected saliva as the specimen — Obtain self-collected saliva sample, perform SARS-CoV-2 testing using the Eppendorf Thermal Cycler Polymerase chain reaction (PCR) system on 30 samples associated with a positive and 30 samples associated with a negative NP sample, then compare saliva results to healthcare worker collected NP sample results evaluated on either the BioFire® FilmArray® Torch® system or the Cepheid® GeneXpert® (gold standard).

SUMMARY:
This is a study that will attempt to validate the process for detecting SARS-CoV-2 (COVID19) on a non-FDA-approved technology using self-collected saliva as the specimen. Investigators will compare self-collected saliva samples and healthcare-worker collected nasopharyngeal samples (Nasal swabs) to see if the self-collected saliva samples are similar in terms of diagnostic accuracy. Investigators will be performing this testing at the site where patients regularly go for COVID19 testing. There will be minimal risk of harm as consenting patients will only have to provide a small amount of saliva into a tube.

DETAILED DESCRIPTION:
This is a descriptive study that will attempt to validate the procedure for detecting SARS-CoV-2 on the Eppendorf Thermal Cycler PCR system using self-collected saliva as the specimen. Investigators will calculate the percent agreement and the 95% confidence intervals (ie, overall agreement, percent positive agreement, and percent negative agreement) between self-collected saliva samples (evaluated on the Eppendorf Thermal Cycler PCR system) and healthcare-worker collected nasopharyngeal samples (evaluated on either the BioFire® FilmArray® Torch® system or the Cepheid® GeneXpert® as the gold standard). Participants without usable results for both the saliva and nasopharyngeal methods will not be included in the analyses. Currently, DGMC uses both FDA Emergency Use Authorization systems interchangeably to test for SARS-CoV-2.

Using human volunteers to obtain positive and negative nasopharyngeal and saliva specimens of SARS-COV-2, this is a test validation study. It uses the Eppendorf Thermal Cycler PCR system to compare the test performance of saliva as a specimen to the standard nasopharyngeal specimen.

This protocol utilizes two different convenience samples of DGMC patients. Patients (i.e. inpatient, outpatients) with a positive COVID-19 test in the past 72 hours, and those who present for COVID-19 testing at DGMC and have negative results. Both groups of patients are willing to provide a saliva sample for COVID-19 testing within 72 hours. The populations will be comprised of active duty, DoD dependents, and retirees who are DGMC patients. This study will enroll at least 60 individuals. Only saliva samples from 30 participants with negative and 30 with positive NP results will be processed. The study will stop recruiting positive patients after obtaining the paired saliva and NP results from 30 participants who are COVID-19 positive by NP test. The study will stop actively recruiting negative patients after obtaining the paired saliva and NP results from 30 participants who are COVID-19 negative by NP test. More than 30 negative patients may be recruited in an attempt to capture 30 positive patients.

Recruitment efforts for positive patients will be conducted utilizing a HIPAA waiver to identify potential study participants, as well as, targeting patients exposed to and/or with symptoms related to COVID-19 who present for COVID-19 testing. The HIPAA Waiver will be used to identify patients (inpatient, outpatient) who have had a positive COVID-19 NP test within the past 72 hours. These patients, as well as others who will have COVID-19 testing at DGMC, will be informed of the study.

Patients interested in participation will make contact with study staff. Those eligible to participate will be given study documents (consent and HIPAA Authorization Form), that will later be reviewed and signed by the patient and study staff. Thereafter, additional information (contact, demographic), and a self-collected saliva specimen will be obtained.

To minimize contact with COVID-19 positive or potentially infected patients when signing documents and obtaining the self-collected saliva sample, staff will wear scrubs (or a lab coat), gloves, eye protection and N95 mask. Documents requiring signature will be signed by the patient while wearing a mask and maintaining a distance of at least 6 feet from study staff or from their vehicle. Consent and HIPAA Authorization Forms will be signed. The original, signed documents will be maintained by study staff and a copy will be provided to the participant. After both documents have been signed, study staff will obtain demographic (age, ethnicity, race and sex) and contact information (name, email address if future contact is desired), date of birth, and the self-collected saliva sample.

Prior to collecting the saliva sample, study staff will ensure the participant has not smoked, eaten or drank anything for the previous 10 minutes. Participants will be given a biohazard bag, label (with a 6-digit numerical code), 25 ml plastic specimen tube without transport medium inside. Then asked to fill it with approximately 2 mL of saliva. There will be a marking on the tube to ensure a sufficient sample is collected. The participant will be instructed to close the lid, place the label on the outside of the tube, then put the labeled tube into the biohazard bag. Participants will then place the bagged specimen inside a second biohazard bag held by either DGMC or a member of the study team. The double-bagged self-collected saliva sample will then be placed into the study cooler containing an ice pack. Saliva specimens will then be transported to the CIF in batch.

After obtaining the paired saliva and NP results from 30 participants who are COVID-19 negative by NP test, saliva testing will only be performed on samples collected from NP positive participants. Patients with unknown COVID-19 status, enrolled in an attempt to capture a COVID-19 positive patient, will have the medical record accessed to retrieve the NP result prior to performing saliva testing. If the NP result is positive, saliva testing will be performed.

Testing will be performed on saliva samples using reverse-transcription polymerase chain reaction (RTPCR). Natural and/or synthetic RNA will be acquired for use as a positive control. RT-PCR will target the E-gene and N-gene of SARS-CoV-2.

1. Within 5 minutes of sample collection the sample will be kept cold for stabilization. A cooler with an ice pack inside will be taken to the location where the participant provides the sample. The sample will be put in a biohazard bag, then immediately be placed into the cooler for transport to the CIF Laboratory in batch.
2. Ribonucleic Acid (RNA) Extraction - Within 12 hours, RNA will be extracted from the specimens using Invitrogen PureLink ® Viral RNA/DNA Mini Kit (Life Technologies). Sample RNA will be stored at -80oC until used.
3. SuperScriptTM III One-Step RT-PCR with PlatinumTM Taq (Life Technologies) will be used for detection and amplification of viral RNA present in specimens using Eppendorf Mastercyler Pro S (Eppendorf). Up to seven primer pairs that are based from CDC and other publications will be used.18-19 Three from the envelope protein gene and four from the nucleocapsid protein gene.
4. Frozen samples will be tested and run in batches.
5. PCR products will be evaluated with gel electrophoresis using the Mini-Protein® Tetra Cell (Bio-Rad).
6. Sequencing - All PCR reactions that produce acceptable amplicons will be stored at -80oC for possible sequencing confirmation using the ABI 3130 (Life Technologies).

Once testing is completed, specimens will be aliquoted and stored at -80oC.

Saliva samples will be interpreted as negative, positive or inconclusive. Negative will be reported when there is no detection in any target; inconclusive when 1 target is detected; and positive when 2 or more targets are detected.

Study staff will access the lab accession number associated with each SARS-CoV-2 positive NP result to request a print out, from the DGMC clinical lab, of the raw data from the instrument used to perform testing. This information will be used to evaluate any discrepancies between the two testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have COVID-19 NP testing at DGMC and are willing to provide a saliva sample within 72 hours
* Adult patients (i.e., inpatient, outpatient) who have positive COVID-19 NP test results at DGMC and are willing to provide a saliva sample within 72 hours of the positive COVID-19 NP test

Exclusion Criteria:

* Patients unwilling to wait or have eaten, drank or smoked within the past 10 minutes
* Patients unwilling or unable to provide 2 mls of saliva
* For positive control participants only, patients whose most recent positive COVID-19 NP test was collected more than 72 hours ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Percent positive agreement between self-collected saliva samples and healthcare-worker collected nasopharyngeal samples | within 1 week of SARS-CoV-2 testing
  Percent positive agreement between self-collected saliva samples (evaluated on the Eppendorf Thermal Cycler PCR system) and healthcare-worker collected nasopharyngeal samples (evaluated on either the BioFire® FilmArray® Torch® system or the Cepheid® GeneXpert® as the gold standard).
Percent negative agreement between self-collected saliva samples and healthcare-worker collected nasopharyngeal samples | within 1 week of SARS-CoV-2 testing
  Percent negative agreement between self-collected saliva samples (evaluated on the Eppendorf Thermal Cycler PCR system) and healthcare-worker collected nasopharyngeal samples (evaluated on either the BioFire® FilmArray® Torch® system or the Cepheid® GeneXpert® as the gold standard).
Percent overall agreement between self-collected saliva samples and healthcare-worker collected nasopharyngeal samples | within 1 week of SARS-CoV-2 testing
  Percent overall agreement between self-collected saliva samples (evaluated on the Eppendorf Thermal Cycler PCR system) and healthcare-worker collected nasopharyngeal samples (evaluated on either the BioFire® FilmArray® Torch® system or the Cepheid® GeneXpert® as the gold standard).

CONTACTS AND LOCATIONS:
Overall Officials: Nolan R Hudson, MS, Principal Investigator — David Grant Medical Center
Locations (1):
- David Grant U.S. Airforce Medical Center, Travis Air Force Base, California, United States

REFERENCES:
- [Background] Fakheran O, Dehghannejad M, Khademi A. Saliva as a diagnostic specimen for detection of SARS-CoV-2 in suspected patients: a scoping review. Infect Dis Poverty. 2020 Jul 22;9(1):100. doi: 10.1186/s40249-020-00728-w. PMID 32698862
- [Background] Azzi L, Carcano G, Gianfagna F, Grossi P, Gasperina DD, Genoni A, Fasano M, Sessa F, Tettamanti L, Carinci F, Maurino V, Rossi A, Tagliabue A, Baj A. Saliva is a reliable tool to detect SARS-CoV-2. J Infect. 2020 Jul;81(1):e45-e50. doi: 10.1016/j.jinf.2020.04.005. Epub 2020 Apr 14. PMID 32298676
- [Background] McCormick-Baw C, Morgan K, Gaffney D, Cazares Y, Jaworski K, Byrd A, Molberg K, Cavuoti D. Saliva as an Alternate Specimen Source for Detection of SARS-CoV-2 in Symptomatic Patients Using Cepheid Xpert Xpress SARS-CoV-2. J Clin Microbiol. 2020 Jul 23;58(8):e01109-20. doi: 10.1128/JCM.01109-20. Print 2020 Jul 23. No abstract available. PMID 32414838
- [Background] Takeuchi Y, Furuchi M, Kamimoto A, Honda K, Matsumura H, Kobayashi R. Saliva-based PCR tests for SARS-CoV-2 detection. J Oral Sci. 2020;62(3):350-351. doi: 10.2334/josnusd.20-0267. PMID 32581183

DOCUMENTS (1):
  • Informed Consent Form (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT04604145/ICF_000.pdf